CLINICAL TRIAL: NCT03798340
Title: Effects of Motor Task-Specific Therapy Synchronized With Vibrotactile Cueing on Sensorimotor Performance of Upper Extremity for the Chronic Stroke Patients
Brief Title: Vibratory Perturbation-based Pinch Task Training for Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-104-206
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Stroke Rehabilitation
Keywords: stroke; perturbation-based training; task-specific motor training; recovery of function
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No

ARMS (2):
- Vibratory perturbed task-specific movement training (Experimental): Intervention: 10 minutes of traditional sensorimotor facilitation followed by 20 minutes of vibratory perturbed task-specific movement training
  Interventions: Other: Vibratory perturbed task-specific movement training; Other: Sensorimotor training
- Traditional task-oriented facilitation (Active Comparator): Intervention:10 minutes of traditional sensorimotor training followed by 20 minutes of reach-to-grasp and hand release training.
  Interventions: Other: Traditional task-oriented facilitation; Other: Sensorimotor training

INTERVENTIONS:
Other: Vibratory perturbed task-specific movement training — The perturbation-based pinch task training was conducted with the affected hand placed on the pinch device. The horizontal vibratory perturbation was generated for a total of 20 minutes by two recoil-type actuators with a frequency of 30 Hz and an amplitude of 2 mm, and intermittent exposure (10 s per 30 s). Each training session was divided into eight cycles with a training interval of 2 min per 2.5 min.
  Arms: Vibratory perturbed task-specific movement training
Other: Traditional task-oriented facilitation — Reach-to-grasp training and hand release training
  Arms: Traditional task-oriented facilitation
Other: Sensorimotor training — Targeted to goals that are relevant to the sensorimotor facilitation of the patient

SUMMARY:
The investigator assumed that perturbed-event-induced vibrotactile cueing enable more precision arm movement adjustment, sensory function and dexterity improvement in the spastic arm. Thus the specific aim of the study was to develop a vibrotactile therapy system that can provide vibrotactile feedback through the pinch performance of the hand when countering mechanically induced perturbations and also analyzed training effects of the perturbation-based pinch task training system on the sensorimotor performance of the hands for stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of unilateral cerebral infarction or hemorrhage
2. Be able to perform a pinch task with the thumb and index finger
3. With premorbid right-handedness

Exclusion Criteria:

1. Subject has a uncontrolled hypertension
2. Subject has major cognitive-perceptual deficits
3. Subject has other brain disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in the result of Fugl-Meyer assessment for UE motor function | baseline, endpoint (6 weeks) and follow up (18 weeks)
  Each item is rated on a three-point ordinal scale (2 points for the detail being performed completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.completely, 1 point for the detail being performed partially, and 0 for the detail not being performed). The maximum motor performance score is 66 points for the upper extremity.
Change in the result of Modified Ashworth scale (MAS) | baseline, endpoint (6 weeks) and follow up (18 weeks)
  Muscle tone is defined by the resistance of a muscle being stretched.The tester graded the resistance felt, with a single score. The higher values represent a worse outcome. 0 point for no increase in muscle tone; 1 point for slight increase in muscle tone, manifested by a catch or by minimal resistance at the end of the range of motion (ROM) when the affected part is moved in flexion or extension; 1 + for slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM; 2 point for more marked increase in muscle tone through most of the ROM, but affected parteasily moved, 3 point for considerable increase in muscle tone and passive movement difficult; 4 point for affected part rigid in flexion or extension.
Change in the result of Box and blocks test | baseline, endpoint (6 weeks) and follow up (18 weeks)
  The score is the number of blocks carried from one box to the other in one minute. Higher values represent a better outcome.
Change in the result of Semmes-Weinstein monofilament (SWM) test | baseline, endpoint (6 weeks) and follow up (18 weeks)
  The Semmes-Weinstein monofilamenttest examines the cutaneous pressure threshold, range from 1.65-6.65. Higher values represent a worse outcome.
Change in the result of Motor Activity Log | baseline, endpoint (6 weeks) and follow up (18 weeks)
  MAL is a structured interview with testing sensitivity used to examine how much (amount of use, AOU) and how well (quality of movement, QOM) the subject uses their more-affected arm. For the 30 items MAL, each item is scored on a 0-5-ordinal scale.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Hsu HY, Kuan TS, Tsai CL, Wu PT, Kuo YL, Su FC, Kuo LC. Effect of a Novel Perturbation-Based Pinch Task Training on Sensorimotor Performance of Upper Extremity for Patients With Chronic Stroke: A Pilot Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 May;102(5):811-818. doi: 10.1016/j.apmr.2020.11.004. Epub 2020 Dec 2. PMID 33278364